CLINICAL TRIAL: NCT02442479
Title: Maximizing Mechanisms of Muscle Hypertrophy to Combat Sarcopenia in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute on Aging (NIA) (NIH); US Dairy Export Council (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5R01AG017896 (NIH)
Record Dates: First submitted 2015-05-06; First posted 2015-05-13 (Estimated); Last update posted 2016-04-25 (Estimated); Status verified 2015-05

CONDITIONS: Aging; Muscular Atrophy
Keywords: exercise; resistance training; muscle strength; muscle hypertrophy
MeSH Terms: conditions — Muscular Atrophy; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- HHH3 (Active Comparator): High-resistance concentric-eccentric training (H) 3 d/wk (HHH3).
  Interventions: Behavioral: resistance training
- HLH3 (Experimental): 3 d/wk mixed model consisting of high-resistance concentric-eccentric training 2 d/wk separated by 1 bout of low-resistance, high-velocity, concentric only training (L) (HLH3).
  Interventions: Behavioral: resistance training
- HH2 (Experimental): High-resistance concentric-eccentric training 2 d/wk (HH2).
  Interventions: Behavioral: resistance training
- HL2 (Experimental): 2 d/wk mixed model consisting of high-resistance concentric-eccentric training 1 d/wk and low-resistance, high-velocity, concentric only training 1 d/wk (HL2).
  Interventions: Behavioral: resistance training

INTERVENTIONS:
Behavioral: resistance training

SUMMARY:
Resistance training has shown the most promise among interventions aimed to combat aging muscle atrophy as it enhances strength, power, and mobility function, but induces varying degrees of skeletal muscle hypertrophy as the investigators demonstrated in the initial 5-year funding period of this award (2001-2006). In the subsequent 5-year funding period (2007-2012), the investigators built on this prior work by using a dose-response approach in older adults - ultimately to optimize the treatment of age-related muscle atrophy. The investigators tested four, long-term resistance training prescriptions in older (60-75 yr) women and men to determine which prescription maximizes mechanisms driving muscle regrowth. One of the innovations in this project was the use of a 4-wk pre-training program to reach a plateau in the early, non-muscle mass adaptations, thereby establishing a true baseline from which both mechanisms of measurable muscle hypertrophy and functional consequences of hypertrophy could be studied in a tightly integrated fashion without bias in the subsequent experimental period. A randomized design was used to test the overarching hypothesis that a novel program of mixed strength and power training would optimize the anabolic environment to promote muscle hypertrophy and robust gains in performance. This hypothesis was tested with three specific aims.

DETAILED DESCRIPTION:
Resistance training has shown the most promise among interventions aimed to combat aging muscle atrophy as it enhances strength, power, and mobility function, but induces varying degrees of skeletal muscle hypertrophy as we demonstrated in the initial 5-year funding period of this award (2001-2006). In the subsequent 5-year funding period (2007-2012), we built on this prior work by using a dose-response approach in older adults - ultimately to optimize the treatment of age-related muscle atrophy. We tested four, long-term resistance training prescriptions in older (60-75 yr) women and men to determine which prescription maximizes mechanisms driving muscle regrowth (protein synthesis and myonuclear addition). One of the innovations in this project was the use of a 4-wk pre-training program to reach a plateau in the early, non-muscle mass adaptations, thereby establishing a true baseline from which both mechanisms of measurable muscle hypertrophy and functional consequences of hypertrophy could be studied in a tightly integrated fashion without bias in the subsequent experimental period. A randomized design was used to test the overarching hypothesis that a novel program of mixed strength and power training would optimize the anabolic environment to promote muscle hypertrophy and robust gains in performance. This hypothesis was tested with three specific aims.

Specific Aim 1. We determined the effects of manipulating intensity, recovery, and mode of contraction on rates of muscle hypertrophy and muscle mass-dependent improvements in tests of in vivo muscle performance among older women and men. In brief, the four training models were: (1) traditional high-resistance concentric-eccentric training (H) 3 d/wk (HHH3); (2) high-resistance concentric-eccentric training 2 d/wk (HH2); (3) 3 d/wk mixed model consisting of high-resistance concentric-eccentric training 2 d/wk separated by 1 bout of low-resistance, high-velocity, concentric only training (L) (HLH3); and (4) 2 d/wk mixed model consisting of high-resistance concentric-eccentric training 1 d/wk and low-resistance, high-velocity, concentric only training 1 d/wk (HL2). For Aim 1, we hypothesized that the HLH3 prescription would prove optimal overall for combined gains in muscle mass, strength, power, and fatigue resistance in both women and men, while HL2 would be the least effective program due to insufficient weekly loading.

Specific Aim 2. Myofiber hypertrophy requires net muscle protein synthesis, and advanced fiber expansion is facilitated by nuclear addition. We are conducting a comprehensive evaluation of: (1) key regulatory steps in the protein synthesis/degradation machinery; and (2) myonuclear addition and satellite cell activation/cell cycle regulation. Quantitative relationships between metabolic/molecular responses and the magnitude of muscle hypertrophy among older adults will enable us to identify underlying factors that respond differently to these four resistance training models, potentially in a gender-specific manner, thus revealing important processes that drive the hypertrophy adaptation. We hypothesized that muscle protein synthesis and myonuclear addition, along with key underlying regulatory processes, would be most favorably affected by the work-recovery cycle of 2 d/wk high-resistance loading (HLH3 and HH2 models), thereby optimizing the anabolic environment for muscle hypertrophy in both older women and men.

Specific Aim 3. To translate the findings under Aim 1 to clinically important outcomes, we determined the degree to which non-traditional resistance training programs lead to improvements in mobility function and weight-bearing exercise difficulty. We hypothesized that a less stressful weekly training regimen consisting of fewer high-resistance contractions (HLH3) and/or fewer training sessions (HH2) while achieving substantial hypertrophy would promote equal or better improvements in mobility function and weight-bearing exercise difficulty than the traditionally prescribed HHH3 program.

ELIGIBILITY:
Inclusion Criteria:

* 60-75 years of age; BMI less than or equal to 30; passed comprehensive physical examination including resting electrocardiogram and a diagnostic graded exercise stress test with 12-lead electrocardiogram; able to exercise on a treadmill for 10 minutes; (female participants) at least 5 years post-menopausal.

Exclusion Criteria:

* Neurological, musculoskeletal, or other disorder that would preclude completing resistance training and all performance tests; uncontrolled hypertension, unstable or exercise-induced angina pectoris or myocardial ischemia; diabetes mellitus; pregnancy; any other medical condition that would interfere with testing or increase one's risk of complications during exercise; lidocaine allergy; prescription anti-coagulants (e.g., Coumadin); current androgen or anabolic (e.g., GH, IGF-I) therapy; food allergy to cow's milk; history of regular resistance exercise during the previous 3 years; any contraindications to magnetic resonance imaging including pacemakers, aneurysm clips, or any other ferrous metal implants; current adherence to a weight reduction diet.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2007-04; Primary Completion 2012-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
muscle mass | Change from baseline at week 35
  DXA-determined lean mass and thigh muscle mass

SECONDARY OUTCOMES:
vastus lateralis muscle fiber size | Change from baseline at week 35
  type I and type II muscle fiber size by immunofluorescence microscopy
maximum strength | Change from baseline at week 35
  one-repetition maximum voluntary strength
maximum power | Change from baseline at week 35
  knee extension power

OTHER OUTCOMES:
sit-to-stand difficulty | Change from baseline at week 35
  relative motor unit activation requirement
steady state exercise difficulty | Change from baseline at week 35
  cardiorespiratory responses to 3 mph walking and 31 steps/min stair climbing
mobility function | Change from baseline at week 35
  6-minute walk test
muscle tissue molecular assays | Change from baseline at week 35
  translation initiation signaling, pro-inflammatory signaling, gene expression

CONTACTS AND LOCATIONS:
Locations (1):
- UAB Center for Exercise Medicine, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Stec MJ, Thalacker-Mercer A, Mayhew DL, Kelly NA, Tuggle SC, Merritt EK, Brown CJ, Windham ST, Dell'Italia LJ, Bickel CS, Roberts BM, Vaughn KM, Isakova-Donahue I, Many GM, Bamman MM. Randomized, four-arm, dose-response clinical trial to optimize resistance exercise training for older adults with age-related muscle atrophy. Exp Gerontol. 2017 Dec 1;99:98-109. doi: 10.1016/j.exger.2017.09.018. Epub 2017 Sep 28. PMID 28964826